CLINICAL TRIAL: NCT01772706
Title: A Randomized, Double Blind, Controlled, Multi-center, Phase III Study to Assess Efficacy of Low Level Diode Laser (100 MW, 658 Nm), in the Prevention and Treatment of Radiochemotherapy-induced Mucositis in Head and Neck Cancer.
Brief Title: Laser Mucite ORL : Effectiveness of Laser Therapy for Mucositis Induced by a Radio-chemotherapy in Head and Neck Cancer
Acronym: LaserMucite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPP400; 2008-003681-26 (EudraCT Number)
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Oral Squamous Cell Carcinoma; Squamous Cell Carcinoma of Oropharynx; Squamous Cell Carcinoma of Hypopharynx; Oral Mucositis
Keywords: Head and neck cancer; Low level laser therapy; Mucositis induced by radiochemotherpy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis; Head and Neck Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- laser low-level energy functional (Experimental): The material used will be a diode laser of 100 mW, with a wavelength of 658 nm. Application will be made after each radiotherapy session in an adapted room (low light intensity, possibility of ENT examination) on all grade superior or equal to 2 stomatitis injuries. The energetic dose delivered will be 4 J/cm2. The duration of the treatment for one will be determined by an abacus.
  Interventions: Procedure: low level laser therapy
- laser low-level energy nonfunctional (Placebo Comparator): The procedure is identical to the one used in arm A but the laser will not be functional. The period of application will be around one minute.
  Interventions: Procedure: placebo (laser low level energy nonfunctional)

INTERVENTIONS:
Procedure: low level laser therapy
  Arms: laser low-level energy functional
Procedure: placebo (laser low level energy nonfunctional)
  Arms: laser low-level energy nonfunctional

SUMMARY:
The purpose of the study is to assess in a randomized, double blind, controlled, multi-center, phase III study, the efficacy of low level diode laser (100 MW, 658 Nm), in the prevention and treatment of radiochemotherapy-induced mucositis for stage III and IV head and neck carcinomas.

DETAILED DESCRIPTION:
This is a Phase III randomized, double-blind, multicenter study, with two groups of patients receiving radiotherapy and concomitant chemotherapy.

The patients will be randomized as follows: Arm A = patients will receive a preventive and curative treatment by low-energy laser, and arm B = a control group treated with standard local treatments and a placebo laser (laser nonfunctional).

Randomization will be balanced in a ratio 1: 1 and stratified by the investigator site. Assessments of mucositis, nutritional status, tolerance of the laser and pain will be performed throughout the treatment, once a week, by an investigator unaware of the patients treatment arm. The locoregional control will be evaluated every 3 months during the first year, then every 6 months up to 5 years. In case of progression, treatments undertaken and their results should be reported.

Radiotherapy: All patients will be treated with conformal radiotherapy with or without IMRT. The dose should be adapted to the treatment indication (exclusive or postoperative) and the histological findings in case of tumoral resection.

The radiotherapy will be prescribed in accordance with the recommendations of the ICRU 50 report. The dose delivered will always be 2 Gy per day 5 times a week. All beams will be treated in each session. A radiological audit will be conducted for each beam treated by photons in the first session and at least once a week.

Chemotherapy:

Several chemotherapies concomitant to radiotherapy are possible:

* a combination of 5-FU and Cisplatin
* a combination of 5-FU and Carboplatin
* Cisplatin alone
* Cetuximab alone

Dental care: All patients (except edentulous) will be seen in odontostomatology consultation prior to the treatment for dental care if necessary or potential production of fluorinated gutters During the treatment, all patients will receive oral care

The dosimetric study will concern the cross section, the frontal and sagittal planes through the axis of the lateral beams.

Arm A : laser low-level energy functional The material used will be a diode laser of 100 mW, with a wavelength of 658 nm. Application will be made after each radiotherapy session in an adapted room (low light intensity, possibility of ENT examination) on all grades superior or equal to 2 stomatitis injuries. The application is painless, athermal, odorless and completely silent. The patient will wear glasses for retinal protection. The operator will also wear glasses for his protection but allowing nevertheless the view of the beams and its limits.

The tumor areas macroscopically invaded will be excluded from the areas application.

The energetic dose delivered will be 4 J/cm2. The duration of the treatment for one will be determined by a corresponding abacus : [t(s) = energy (J/cm2) x surface (cm2) / puissance (W)]. The overall duration will be a few minutes varying depending on the surface to be treated The usual dental care will be prescribed when required.

Arm B : laser low-level energy nonfunctional The procedure is identical to the one used in arm A but the laser will not be functional. The period of application will be around one minute. All applications will be performed by one single operator by center. The results will be assessed once a week by another physician (or nurse specifically trained) in each center, unaware of whether the patients had laser sessions or not, in order to respect the "blinding". The assessment will be detailed on a specifique sheet, specifying the degree of mucositis (WHO), the level of pain, body weight , type of feeding , any analgesic treatment taken by the patient, quality of life specific questionnaire, and the possible end of treatment or therapeutic modifications (number of cycles of chemotherapy, dosage).

The laser should be started as soon as a grade 2 mucositis (WHO) is observed and will be continued throughout the radio-chemotherapy until improvement of the mucositis (grade <2).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Patient with squamous cell carcinoma of the oral cavity, oropharynx or hypopharynx, stage III-IV, histologically confirmed
3. PS > or = 2
4. Estimated life expectancy greater than 3 months in the absence of treatment
5. Concomitant chemotherapy with one of the following choices not prohibited:

   * Cetuximab alone
   * 5-FU combined to Carboplatin or Cisplatin
   * Cisplatin alone Being defined as follows: serum creatinine < 150 µmol/l and creatinine clearance superior or equal to 55ml/min (calculated with the Cockcroft method) in case of serum creatinine > 120 µmol/l
6. Appropriate hematological, renal and hepatic function parameters, within 15 days prior to randomization, with the following results:

   * Hemoglobin> 8g/dL
   * Neutrophils> 1500 x 109 / L
   * Platelets> 100 x 109 / l
   * Total bilirubin <1.5 times the upper limit of normal
   * ALT / AST and alkaline phosphatase <2.5 times the upper limit of normal.
7. For women of childbearing potential, a reliable contraceptive measure (hormonal contraception, intrauterine device) is required.

Exclusion Criteria:

1. Presence of other malignancies either concomitant or diagnosed within the last five years, except basal cell carcinoma or in situ carcinoma of the cervix
2. Neoadjuvant chemotherapy
3. Metastatic disease
4. Previous treatment with ENT radiotherapy
5. Severe hypersensitivity known to platinum based agent
6. Any uncontrolled pathology (respiratory, cardiac, hepatic or renal)
7. Pregnant or breastfeeding women (a seric or urinary pregnancy test must be negative at the time of study entry for women of childbearing age).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-10-30 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of preventive and curative low energy laser induced mucositis in patients receiving concomitant chemotherapy and radiotherapy for squamous cell carcinoma of the head and neck with stage III-IV | 7 weeks

SECONDARY OUTCOMES:
To evaluate the pain by a numerical analog, in its the nature and the dosage of analgesics consumed. | 7 weeks
To assess the nutritional status by body weight follow-up and the capability of swallowing various foods, and biologically the serum albumin, prealbumin, and optionally a measure of body fat (impedance, skinfolds) | 7 weeks
To assess the treatment compliance by the spread and discontinuation of radiation therapy, in duration (days) and the cause of discontinuations, the number of cycles of chemotherapy administered, and dose modifications or possible delays. | 7 weeks
To assess the laser tolerance | 7 weeks
To assess the quality of life using the QLQ-HN35 questionnaire. | 7 weeks

OTHER OUTCOMES:
To evaluate the Locoregional control every 3 months for 1 year, then every 6 months up to 5 years. | 5 years
To calculate the Disease-free survival from the date of randomization to the first event (recurrence or death) or up to 5 years. | 5 years
To document the Overall survival calculated from the date of randomization to death from any cause or up to 5 years. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric JADAUD, MD, Principal Investigator — Institut de Cancerologie de l'Ouest - Paul Papin
Locations (6):
- France (6):
  - Institut de Cancerologie de l'Ouest Paul Papin, Angers
  - Centre Guillaume le Conquérant, Le Havre
  - Hôpital La Pitié Salpêtrière, Paris
  - Centre hospitalier universitaire La Milétrie, Poitiers
  - Centre Jean Godinot, Reims
  - Clinique Armoricaine de Radiologie, Saint-Brieuc

REFERENCES:
- [Derived] Legoute F, Bensadoun RJ, Seegers V, Pointreau Y, Caron D, Lang P, Prevost A, Martin L, Schick U, Morvant B, Capitain O, Calais G, Jadaud E. Low-level laser therapy in treatment of chemoradiotherapy-induced mucositis in head and neck cancer: results of a randomised, triple blind, multicentre phase III trial. Radiat Oncol. 2019 May 22;14(1):83. doi: 10.1186/s13014-019-1292-2. PMID 31118057